CLINICAL TRIAL: NCT06404827
Title: Investıgatıon of the Effect of Hıppotherapy Sımulator on Lower Extremıty Selectıve Motor Control, Balance and Trunk Control in Chıldren Wıth Spastıc Cerebral Palsy
Brief Title: The Effect of Hippotherapy Simulator in Children with Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Yalcın KARABULUT, Principal investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKU-FTR-YK-1
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Horseback riding simulator; Selective motor control; Balance
MeSH Terms: conditions — Cerebral Palsy | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Horseback riding simulator+Routine physiotherapy) (Experimental): Horseback riding simulator (HRS) will be applied in addition to routine Physiotherapy and Rehabilitation. This group will receive 20 minutes of routine physiotherapy training and 20 minutes of HRS application in addition to 2 sessions per week for 8 weeks.
  Interventions: Other: Horseback riding simulator; Other: Routine Physiotherapy and Rehabilitation
- Control group (Routine physiotherapy) (Active Comparator): Routine physiotherapy training will be applied within a specific programme for 40 minutes in 2 sessions per week for 8 weeks.
  Interventions: Other: Routine Physiotherapy and Rehabilitation

INTERVENTIONS:
Other: Horseback riding simulator — Horseback riding simulator (HRS) will be applied in addition to routine Physiotherapy and Rehabilitation.
  Arms: Intervention group (Horseback riding simulator+Routine physiotherapy)
Other: Routine Physiotherapy and Rehabilitation — Routine Physiotherapy and Rehabilitation within a spesific programme

SUMMARY:
The horseback riding simulator (HRS) is a dynamic robotic device that mimics the movement of a horse for hippotherapy purposes. HRS aims to improve the patient's balance, adaptation and provide postural adjustment by mimicking the rhythmic movements of the horse.

This study aims to research the potential benefits of the horseback riding simulator on the lower extremity selective motor control, balance and trunk control in children with Cerebral palsy.

DETAILED DESCRIPTION:
Between the dates of the study, children with Cerebral palsy (CP) who meet the inclusion criteria will be allocated into two groups (intervention group, control group) by randomiZation method.

Intervention group: horseback riding simulator (HRS) will be applied in addition to routine Physiotherapy and Rehabilitation. This group will receive 20 minutes of routine physiotherapy training and 20 minutes of HRS application in addition to 2 sessions per week for 8 weeks.

Control group: Routine physiotherapy training will be applied within a specific programme for 40 minutes in 2 sessions per week for 8 weeks.

All the assessments will be performed before and after the training in the 8-week groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Spastic Cerebral Palsy
* Voluntary participation
* Age between 5-17 years,
* GMFCS Level I-II-III
* MACS Level I-II-III
* Modified Asworth Scale (MAS) Level 1-2-3
* Have the ability to sit with support

Exclusion Criteria:

* Having severe visual and hearing problems
* Severe distractibility problems and inability to follow task instructions,
* Not voluntary to participate in the research,
* Individuals with CP who have had hip or spine surgery in the last 6 months
* Individuals with CP who have undergone Botox in the last 6 months

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | At Baseline
  Assessing functional level and gross motor function of children with CP. Level I refers to a child walking independently, while level V refers to mobility with a wheelchair.
Manuel ability classification system (MACS) | At Baseline
  Classify how children with CP use their hands when dealing with objects in daily activities. It is a 5-level classification scale. The higher the level, the worse the manual ability. Level 1 means that objects can be handled and used easily and successfully. Level 5 refers to being unable to handle and use objects and having severely limited ability to perform even simple activities.
Change from Baseline Selective Control Assessment of the Lower Extremity at 8 weeks | Change from Baseline at 8 weeks
  Evaluates the lower extremity selective motor control of individuals with CP. The scale assesses five joints separately and bilaterally: hip, knee, ankle, subtalar joint and toe. The degree of selective motor control is determined for each joint as 'normal' (2 points), 'impaired' (1 point) or 'unable to perform' (0 points), according to the patient's ability to perform the movements. The total score is obtained by summing the scores from the joint levels for each limb, with a maximum score of 10 points. Low scores indicate poor selective motor control.
Change from Baseline Pediatric balance scale at 8 weeks | Change from Baseline at 8 weeks
  Assesses the balance of children with CP. This scale consists of 14 items, each of which is scored from 0 to 4. A score of 0 indicates that he/she cannot carry out the instruction and a score of 4 indicates that he/she can do it without difficulty. The total score ranges from 0-56. A low total score indicates a decrease in balance function.
Change from Baseline Trunk Control Measurement Scale at 8 weeks | Change from Baseline at 8 weeks
  This scale consists of two main parts, dynamic and static sitting balance, and provides an assessment. The scale consists of 15 items. Items are scored as 0, 1, 2 or 3. The minimum score that can be obtained from the scale is 0 and the maximum score is 58. A higher score indicates better trunk control.
Change from Baseline Modified Ashworth Scale (MAS) at 8 weeks | Change from Baseline at 8 weeks
  This scale is the most widely used clinical scale to assess spasticity. It is a 6-point scale that assesses muscle tone by passively moving the joint through the normal range of possible motion and recording resistance to passive movement. The scoring ranges from 0-5. There is no tonus increase at 0. 5 indicates that the affected limb is rigid. The higher the score, the greater the increase in tonus.

CONTACTS AND LOCATIONS:
Overall Officials: Yalçın Karabulut, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No